CLINICAL TRIAL: NCT04706247
Title: Segmental High Thoracic Combined Spinal Epidural Anesthesia for Breast Surgery
Brief Title: Thoracic Combined Spinal Epidural Anesthesia for Breast Surgery
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: lutfi1
Record Dates: First submitted 2021-01-10; First posted 2021-01-12 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-01

CONDITIONS: Pain; Breast Diseases
MeSH Terms: conditions — Pain; Breast Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: thoracic combined spinal epidural anesthesia — A combined spinal-epidural anesthesia set will be used for the block. Using the loss of resistance to saline technique, an 18 G Tuohy needle will be advanced to the T2-3 vertebral interspace with the mid-line approach. After confirming the epidural space, a 26 G pencil point spinal needle will be inserted slowly through the Tuohy needle to puncture the dura. After free flow of cerebrospinal fluid will be observed, local anesthetic wil be injected into the subarachnoid space over 15 secs. Then, an epidural catheter will be inserted into the epidural space.

SUMMARY:
The aim of the study is to investigate the efficacy of the thoracic combined spinal epidural anesthesia in breast surgery.

DETAILED DESCRIPTION:
Previous studies of the regional anesthetic techniques such as erector spinae plane block and pectoralis nerve blocks (PECs blocks) additional to general anesthesia have described their use for postoperative analgesia in breast surgery. It has been also reported that these blocks can be used to provide surgical anesthesia in breast surgery . Segmental thoracic epidural anesthesia can be used as an alternative anesthetic technique in patients with severe chronic obstructive pulmonary disease and asthma undergoing breast surgery. It has been also reported that thoracic spinal anesthesia was effective and successful in patients undergoing laparoscopic surgery. In this study, efficacy of high thoracic spinal epidural anesthesia in patients undergoing breast surgery will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be to undergo elective surgery for breast surgery
* American Society of Anesthesiologists (ASA) physical status classification groups I or II

Exclusion Criteria:

* body mass index>35 kg/m2,
* presence of any condition complicating and contraindicating spinal epidural anesthesia.

Ages: 18 Months to 70 Months | Sex: Female
Age Groups: Child
Study Population: Adults between 18-75 years of age and who will be to undergo elective breast surgery
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Block success | through study completion, an average of 3 months
  the number of patients whose surgery was completed without general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Lutfi Ozyurek, M.D., Study Director — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)